CLINICAL TRIAL: NCT01804348
Title: AL-SENSE 1-Step - Determination of Product Specificity
Acronym: ROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Common Sense (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: F-7-32.2-1; 0096-12-NHR (Registry Identifier: Helsinky committee)
Record Dates: First submitted 2013-02-19; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2012-11

CONDITIONS: PREMATURE RUPTURE OF MEMBRANES
Keywords: PROM
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL-SENSE 1-Step (Experimental): a single AL-SENSE 1-Step to use up to 12 hours or until they notice any wetness.
  Interventions: Device: AL-SENSE 1-Step

INTERVENTIONS:
Device: AL-SENSE 1-Step — a single AL-SENSE 1-Step to use up to 12 hours or until they notice any wetness.

SUMMARY:
Clinical diagnosis of amniotic fluid leak will be determined, according the hospital standard procedure, using pooling test and/or sterile speculum examination and /or pH test, and AmniSure, N-Dia, Inc. (immunoassay for diagnosis of ruptured fetal membranes (ROM)). Amniotic fluid leak test, using the AL- SENSE 1-Step device, will be considered positive in case of presence of a blue or green or grey stain on a yellow background of the AL-SENSE 1-Step, as observed by the patient and the clinician (positive/negative).

DETAILED DESCRIPTION:
Pregnant women arriving at the hospital and reporting unidentified wetness (undetermined whether they sense amniotic fluid leakage or urinary incontinence) will receive a single AL-SENSE 1-Step to use up to 12 hours or until they notice any wetness. The clinician will explain the proper use and handling of the AL-SENSE 1-Step and how to read the result.

In each case, the subject and the clinician/midwife (non bias to the hospital standard procedure results) will be required to read and record any occurrence of color change of the AL-SENSE 1-Step immediately after removing the test to mark if it changes color to blue or to green or to grey on the designated form.

The non bias physician, who is not aware to the AL-SENSE 1-Step result (other than the clinician/midwife who records the AL-SENSE 1-Step results) will perform a diagnosis tests for amniotic fluid leak detection, according to the hospital standard procedure.

The investigator will compare the AL-SENSE 1-Step results reading of the patient to the clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. AgE 18 years OR GREATER.
2. Subject who will sign the informed consent form.
3. Subject who arrive at the obstetric department reporting a feeling of vaginal wetness feeling (undetermined whether she sense amniotic fluid leakage or urinary incontinence).

Exclusion Criteria:

1. Subjects that have had sexual relations within the last 12 hours.
2. Subject is unable or unwilling to cooperate with study procedures.
3. Subject is currently participating in another clinical study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
amniotic fluid leaks | up to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstain, MD, Principal Investigator — Western Galilee Hospital Nahariya, Israel
Locations (1):
- Western Galilee Hospital, Nahariya, Israel